CLINICAL TRIAL: NCT05684120
Title: Mood Lifters for Undergraduates Project
Brief Title: Mood Lifters for Undergraduates
Acronym: ML-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Patricia Deldin, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00221612
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Depression; Anxiety; Mood Disorders; Mental Health Wellness 1; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Waitlist control model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Individuals in this arm will take part in the Mood Lifters program immediately after recruitment.
  Interventions: Behavioral: Mood Lifters for Undergraduates
- Waitlist Control Group (No Intervention): Individuals in this arm will be invited to take part in the Mood Lifters program after they complete post-treatment surveys as part of the control group.

INTERVENTIONS:
Behavioral: Mood Lifters for Undergraduates — Participants will need to attend 14 hour-long virtual weekly meetings on Zoom that focus on helpful mental health strategies and skills. Participants will be encourage to practice what they learn at home in order to improve their mood or mental wellness.
  Other Names: Mood Lifters for College Students
  Arms: Treatment Group

SUMMARY:
Large-scale, effective, low-cost, and evidence-based programs that can nimbly translate new research discoveries into prevention and care for psychosocial-based problems are urgently needed since the vast majority of people who need evidence-based care do not receive it.

The purpose of this randomized control trial is to investigate the feasibility and efficacy of a Mood Lifters group template specifically for undergraduate students. Mood Lifters is an effective peer-led program that improves or maintains mental health. It seeks to help people enhance pleasure, engagement, and meaning in their lives while minimizing depression, fear, loneliness, and other negative feelings via a proprietary peer-based program that offers weekly meetings and other flexible support options. One obstacle to providing mental health care in the US is that it is costly to provide one-on-one therapy by a licensed professional. This is particularly true in large group settings with limited resources (counseling centers) and a large need for mental health care, like universities.

ELIGIBILITY:
Inclusion:

* undergraduate students
* at least 18 years of age

Exclusion criteria include:

* active suicidal thoughts or behavior
* active psychosis
* borderline personality disorder
* active mania
* unwillingness to attend all sessions or treatment types (e.g., unwillingness to attend remote)
* non-undergraduate students.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-18 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 | through study completion, an average of 1 year
  Assesses Depressive Symptoms (Range 0-27; higher scores indicate more significant symptoms of depression)
Generalized Anxiety Disorder - 7 | through study completion, an average of 1 year
  Assesses Anxiety Symptoms (Range 0-21; higher scores indicate more significant symptoms of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Deldin, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No